CLINICAL TRIAL: NCT06474065
Title: Pregnancy Outcomes Following Hysteroscopic, Laparoscopic and Laparotomic Myomectomy
Brief Title: Pregnancy Outcomes Following Myomectomy
Status: Completed | Type: Observational
Sponsor: Centro di Ricerca Clinica Salentino (Network)
Responsible Party: Sponsor
Other Study IDs: CER 0324
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Uterine Fibroid; Pregnancy Complications; Reproductive Issues; Reproductive Sterility
Keywords: Fibroids; Leiomyoma; Myomectomy; Outcome; Pregnancy
MeSH Terms: conditions — Leiomyoma; Pregnancy Complications; Infertility | interventions — Uterine Myomectomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treated patiens' Group as Group 1: Patients submitted to hysteroscopic, laparoscopic or laparotomic myomectomy
  Interventions: Procedure: Myomectomy
- Untreated patiens' Group as Group 2: Control group - unoperated patients

INTERVENTIONS:
Procedure: Myomectomy — Patients submitted to operation of fibroids removal
  Groups: Treated patiens' Group as Group 1

SUMMARY:
The most prevalent genital pathology, uterine fibroids have a detrimental impact on the health of women. Fibroid symptoms are typically more impactful on females and frequently require uterine excision. Although contentious in terms of how it affects pregnancy outcomes, hysteroscopic, laparoscopic, or laparotomic myomectomy has always been a necessary and suitable procedure for the patient's health. Numerous studies have been conducted on the topic, but no clear findings have been reached.

The goal of this observational study is to investigate the pregnancy outcomes after hysteroscopic, laparoscopic, laparotomic myomectomies in female patients affected by fibroids. The main questions it aims to answer are:

To investigate pregnancy outcomes in relation to surgical approach used for myomectomy.

To investigate whether pregnancy outcome is different in relation to time when myomectomy was performed: on a pregnant uterus or on a non-gravid uterus.

If there is a comparison group: Researchers will compare a group of patients unsubmitted to surgery, to see the difference with the operated patients.

Participants will follow up, to evaluate the possible pregnancy complications, the intraoperative complications and other perinatal and post-operative complications.

DETAILED DESCRIPTION:
AIMS:

1. To investigate pregnancy outcomes in relation to surgical approach used for myomectomy.
2. To investigate if pregnancy outcome is different in relation to time when myomectomy was performed: on a gravid uterus or on a non-gravid uterus

Patients enrolled are divided in three major groups:

* Group A: myomectomy outside of pregnancy-A1 hysteroscopic; A2 laparoscopic; A3 laparotomy
* Group B: myomectomy during CS: B1 trans-endometrial; B2 serosal
* Group C: control group with repeated CS

INCLUSION CRITERIA:

1. women of reproductive age (up to 45 yrs)-all groups
2. women who had myomectomy (group A and B)/CS (group C) at least two years before the enrolment
3. myomas 30 mm in size and larger (groups A and B)
4. Study groups: myomectomy performed as hysteroscopic/laparoscopic/laparotomic myomectomy or cesarean myomectomy, both using transendometrial or serosal approach: gravida 2 para 2 or gravida 1 para 1 [groups A1, A2, A3 and groups B1 and B2]
5. Control group: women who had cesarean section in their second pregnancy-para 2 gravida 2, at least two years after the CS [group C]

EXCLUSION CRITERIA:

1. any previous surgery on reproductive organs except myomectomy
2. any additional operation during cesarean myomectomy procedure except cesarean section
3. history of endometriosis or PID
4. coagulation disorders
5. previous treatment for any malignant disease
6. previous GTD
7. premature ovarian failure or any kind of ovarian insufficiency necessitating oocyte donation
8. systemic diseases: IBD, MS, DM

DATA TO COLLECT:

1. age
2. years after myomectomy or CS(for group C)
3. gravidity
4. parity
5. BMI
6. myoma characteristics (size and type)
7. myomectomy procedure
8. gestational week at delivery
9. primary indication for CS
10. fetal position
11. placental pathology
12. preoperative hematologic values
13. postoperative hematologic values
14. duration of the CS
15. myoma recurrence in groups A and B
16. uterine rupture
17. perioperative transfusion
18. febrile morbidity
19. postoperative hospitalization in days
20. PPH
21. cause of PPH
22. uterine atony
23. relaparotomy
24. hysterectomy
25. blood vessels ligation
26. fetal presentation: cephalic/other
27. neonatal body weight
28. Apgar score

OUTCOMES:

1. pregnancy complications

   1. placental pathology: placenta previa, placental abruption, PAS
   2. PPROM (gestational age)
   3. abnormal presentation: cephalic/other
   4. uterine rupture: complete/incomplete
   5. preterm/term delivery (gestational age at delivery)
2. intraoperative complications

   1. intraabdominal adhesions/PAI score
   2. surgery complications: Claven Dindo classification
3. other complications:

   1. neonatal outcome,
   2. duration of maternal hospitalization,
   3. primary or secondary PPH
   4. primary or secondary PPH
   5. relaparotomy
   6. peripartum hysterectomy,
   7. ligation of major blood vessels (uterine, ovarian, iliac)

The study will be conducted as a multicentric observational study including cesarean section deliveries in each participating center. In each participating center, one person will be in charge for data collection and filling the SPSS database after obtaining the approval of the local Ethic Committee. As the study is observational and all the procedures will be conducted according to the local practice, informed consent from patients is not necessary.

Following data collection and termination of the study, a single researcher will oversee the SPSS data collection for all the participating centers, checking the quality of data and submitting it for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. women of reproductive age (up to 45 yrs)-all groups
2. women who had myomectomy (group A and B)/CS (group C) at least two years before the enrolment
3. myomas 30 mm in size and larger (groups A and B)
4. Study groups: myomectomy performed as hysteroscopic/laparoscopic/laparotomic myomectomy or cesarean myomectomy, both using transendometrial or serosal approach: gravida 2 para 2 or gravida 1 para 1 [groups A1, A2, A3 and groups B1 and B2]
5. Control group: women who had cesarean section in their second pregnancy-para 2 gravida 2, at least two years after the CS [group C]

Exclusion Criteria:

1. any previous surgery on reproductive organs except myomectomy
2. any additional operation during cesarean myomectomy procedure except cesarean section
3. history of endometriosis or PID
4. coagulation disorders
5. previous treatment for any malignant disease
6. previous GTD
7. premature ovarian failure or any kind of ovarian insufficiency necessitating oocyte donation
8. systemic diseases: IBD, MS, DM

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients to submit to myoemctomy, are divided in three major groups:
  * Group A: myomectomy outside of pregnancy-A1 hysteroscopic; A2 laparoscopic; A3 laparotomy
  * Group B: myomectomy during CS: B1 trans-endometrial; B2 serosal
  * Group C: control group with repeated CS
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2024-06-28 (Actual); Primary Completion 2025-10-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Pregnancy complications | 1 year
  placental pathology, intraoperative complications, other complications

SECONDARY OUTCOMES:
Intraoperative complications | 1 year
  intraabdominal adhesions/PAI score, surgical complications: Claven Dindo classification

OTHER OUTCOMES:
other complications | 1 year
  neonatal outcome, duration of maternal hospitalization, Primary or secondary PPH, relaparotomy, peripartum hysterectomy, ligation of major blood vessels

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Tinelli, MD, Principal Investigator — Centro di Ricerca Clinica Salentino
Locations (1):
- Andrea Tinelli, Lecce, Le, Italy

IPD SHARING:
Plan to Share IPD: Yes
I am considering making individual participant data (IPD) available to other researchers.
Supporting Information: Study Protocol
Time Frame: 1 year
Access Criteria: I'm considering to make IPD Sharing Access Criteria

REFERENCES:
- [Result] Hatirnaz S, Guler O, Basbug A, Cetinkaya MB, Kanat-Pektas M, Bakay K, Celik S, Senturk S, Soyer-Caliskan C, Gurcaglar A, Sahin B, Kalkan U, Celik H, Kalyoncu S, Biyik I, Yassa M, Erol O, Akarsu S, Turhan U, Ulubasoglu H, Sparic R, Tinelli A. A Comparative Multicentric Study on Serosal and Endometrial Myomectomy During Cesarean Section: Surgical Outcomes. J Invest Surg. 2021 Jul;34(7):687-694. doi: 10.1080/08941939.2020.1725188. Epub 2020 Feb 17. PMID 32064967
- [Result] Sparic R, Andric L, Guler O, Malvasi A, Babovic I, Hatirnaz S, Dellino M, Tinelli A. Cesarean Myomectomy: Reflections on Clinical and Surgical Controversies between a New Trans-Decidual Technique vs. Traditional Method. Medicina (Kaunas). 2024 Apr 8;60(4):609. doi: 10.3390/medicina60040609. PMID 38674255
- [Result] Hatirnaz S, Guler O, Basaranoglu S, Tokgoz C, Kilic GS. Endometrial myomectomy: a novel surgical method during cesarean section. J Matern Fetal Neonatal Med. 2018 Feb;31(4):433-438. doi: 10.1080/14767058.2017.1286320. Epub 2017 Feb 9. PMID 28114870
- [Result] Tinelli A, Kosmas I, Medvediev MV, Malvasi A, Morciano A, Sparic R, Mynbaev OA. Myomectomy in adult women of reproductive age: a propensity score-matched study for pregnancy rates. Arch Gynecol Obstet. 2023 Oct;308(4):1351-1360. doi: 10.1007/s00404-023-07135-0. Epub 2023 Jul 14. PMID 37450263
- [Result] Tinelli A, Hurst BS, Hudelist G, Tsin DA, Stark M, Mettler L, Guido M, Malvasi A. Laparoscopic myomectomy focusing on the myoma pseudocapsule: technical and outcome reports. Hum Reprod. 2012 Feb;27(2):427-35. doi: 10.1093/humrep/der369. Epub 2011 Nov 16. PMID 22095838
- [Result] Sparic R, Papoutsis D, Bukumiric Z, Kadija S, Spremovic Radjenovic S, Malvasi A, Lackovic M, Tinelli A. The incidence of and risk factors for complications when removing a single uterine fibroid during cesarean section: a retrospective study with use of two comparison groups. J Matern Fetal Neonatal Med. 2020 Oct;33(19):3258-3265. doi: 10.1080/14767058.2019.1570124. Epub 2019 Jan 30. PMID 30700185
- [Result] Tinelli A, Malvasi A, Mynbaev OA, Barbera A, Perrone E, Guido M, Kosmas I, Stark M. The surgical outcome of intracapsular cesarean myomectomy. A match control study. J Matern Fetal Neonatal Med. 2014 Jan;27(1):66-71. doi: 10.3109/14767058.2013.804052. Epub 2013 Jun 20. PMID 23662726
- [Result] Sparic R, Malvasi A, Kadija S, Stefanovic A, Radjenovic SS, Popovic J, Pavic A, Tinelli A. Safety of cesarean myomectomy in women with single anterior wall and lower uterine segment myomas. J Matern Fetal Neonatal Med. 2018 Aug;31(15):1972-1975. doi: 10.1080/14767058.2017.1333096. Epub 2017 Jun 6. PMID 28585458
- [Result] Tinelli A, Favilli A, Lasmar RB, Mazzon I, Gerli S, Xue X, Malvasi A. The importance of pseudocapsule preservation during hysteroscopic myomectomy. Eur J Obstet Gynecol Reprod Biol. 2019 Dec;243:179-184. doi: 10.1016/j.ejogrb.2019.09.008. Epub 2019 Sep 17. PMID 31585677
- [Result] Tinelli A, Malvasi A, Hurst BS, Tsin DA, Davila F, Dominguez G, Dell'edera D, Cavallotti C, Negro R, Gustapane S, Teigland CM, Mettler L. Surgical management of neurovascular bundle in uterine fibroid pseudocapsule. JSLS. 2012 Jan-Mar;16(1):119-29. doi: 10.4293/108680812X13291597716302. PMID 22906340
- [Result] Tinelli A, Mettler L, Malvasi A, Hurst B, Catherino W, Mynbaev OA, Guido M, Alkatout I, Schollmeyer T. Impact of surgical approach on blood loss during intracapsular myomectomy. Minim Invasive Ther Allied Technol. 2014 Mar;23(2):87-95. doi: 10.3109/13645706.2013.839951. Epub 2013 Sep 18. PMID 24044380
- [Result] Mettler L, Schollmeyer T, Tinelli A, Malvasi A, Alkatout I. Complications of Uterine Fibroids and Their Management, Surgical Management of Fibroids, Laparoscopy and Hysteroscopy versus Hysterectomy, Haemorrhage, Adhesions, and Complications. Obstet Gynecol Int. 2012;2012:791248. doi: 10.1155/2012/791248. Epub 2012 Apr 9. PMID 22619681
- [Result] Tinelli A, Malvasi A, Hudelist G, Cavallotti C, Tsin DA, Schollmeyer T, Bojahr B, Mettler L. Laparoscopic intracapsular myomectomy: comparison of single versus multiple fibroids removal. An institutional experience. J Laparoendosc Adv Surg Tech A. 2010 Oct;20(8):705-11. doi: 10.1089/lap.2010.0082. PMID 20701546